CLINICAL TRIAL: NCT06251947
Title: A Study of Efbemalenograstim Alfa Injection for Ovarian or Cervical Cancer Receiving Chemotherapy Regimen With Risk Factors:A Single-Arm, Multicenter Clinical Trial
Brief Title: Efbemalenograstim Alfa Injection for Ovarian or Cervical Cancer Receiving Chemotherapy Regimen
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Beihua Kong, Clinical Professor, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Guard-05; Guard-05 (Other: Chia Tai Tianqing Pharmaceutical Group Co., Ltd.)
Record Dates: First submitted 2024-01-22; First posted 2024-02-09 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Cancer; Cervical Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Efbemalenograstim Alfa should be administered subcutaneously, 20mg per injection, within 24-48 hours after the completion of each chemotherapy cycle.
  Interventions: Drug: Efbemalenograstim Alfa

INTERVENTIONS:
Drug: Efbemalenograstim Alfa — Efbemalenograstim Alfa is indicated to decrease the incidence of infection, as manifested by febrile neutropenia, in adult patients with non-myeloid malignancies receiving myelosuppressive anti-cancer drugs associated with a clinically significant incidence of febrile neutropenia.

SUMMARY:
The aim of this study was to observe the efficacy and safety of Efbemalenograstim Alfa in the prevention of absolute neutrophil count (ANC) reduction after chemotherapy in Ovarian and Cervical cancer patients at risk of platinum-containing chemotherapy with risk factors in febrile neutropenia (FN).

DETAILED DESCRIPTION:
This study is a single-arm, multicenter clinical trial. A total of 83 patients will be enrolled, including 55 patients with primary epithelial ovarian cancer (including fallopian tube cancer and primary peritoneal cancer) and 28 patients with primary or recurrent/metastatic cervical cancer in the first-line setting.

1) Ovarian Cancer

Chemotherapy regimen (Paclitaxel + Carboplatin ± Bevacizumab):

Paclitaxel 175mg/m2, intravenous infusion over 3 hours, on day 1; followed by Carboplatin Area under the curve 5(AUC5), intravenous infusion over 1 hour, on day 1; Bevacizumab 7.5-15 mg/kg, on day 1, administered as intravenous infusion; repeated every 3 weeks.

(2) Cervical Cancer

Chemotherapy regimen (Paclitaxel + Carboplatin/Cisplatin ± Bevacizumab):

Paclitaxel 175mg/m2, intravenous infusion over 3 hours, on day 1; followed by Carboplatin AUC5, intravenous infusion over 1 hour, on day 1, or Cisplatin 50-80mg/m2, intravenous infusion over 1-3 hours, on day 1; Bevacizumab 7.5-15 mg/kg, on day 1, administered as intravenous infusion; repeated every 3 weeks.

Efbemalenograstim Alfa should be administered subcutaneously, 20mg per injection, within 24-48 hours after the completion of each chemotherapy cycle.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old and ≤ 70 years old.
2. First-line epithelial ovarian cancer (including fallopian tube cancer and primary peritoneal cancer) and first-line treatment or recurrent/metastatic cervical cancer.
3. Planned to receive 3-6 cycles of paclitaxel + carboplatin/cisplatin ± bevacizumab therapy.
4. Eastern Cooperative Oncology Group (ECOG) score < 2.
5. Expected survival time > 3 months.
6. Before enrollment, neutrophil count (ANC) ≥ 2.0 × 10^9/L, hemoglobin (Hb) ≥ 90.0 g/L, and platelet (PLT) ≥ 80 × 10^9/L.
7. Associated with ≥ 1 self-factors increasing the risk of febrile neutropenia (FN): ① age > 65 years, receiving full-dose intensity chemotherapy; ② history of previous chemotherapy or radiotherapy; ③ persistent neutropenia; ④ tumor involvement of the bone marrow; ⑤ recent surgery and/or open wounds; ⑥ hepatic dysfunction (bilirubin > 2.0 mg•dL-1); ⑦ renal dysfunction (creatinine clearance rate < 50 mL•min-1); ⑧ history of previous FN occurrence; ⑨ concomitant malignant hematological or lymphatic system diseases; ⑩ chronic immunosuppression; ⑪ poor nutritional/physical status. Individualized judgment and decision-making based on the patient's specific condition are required in clinical practice.
8. Left ventricular ejection fraction (LVEF) > 50%.
9. Women who are not capable of reproduction, i.e., postmenopausal for at least 1 year or have undergone sterilization procedures (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy). Fertile patients agree to use appropriate contraceptive measures within 1 month before the start of the trial and up to 30 days after the end of the study, such as condoms, spermicidal condoms, foam, gel, diaphragm, intrauterine device (IUD), contraceptive pills (oral or injectable), etc.
10. Willing to provide written informed consent and to compliant study procedure.
11. The investigator determines that the patient can tolerate treatment with Efgbemalenograstim alfa.

Exclusion Criteria:

1. Uncontrolled infection or systemic antibiotic therapy within 72 hours prior to chemotherapy.
2. Pregnant or lactating women.
3. History of bone marrow or stem cell transplantation.
4. Concurrent malignancies other than primary ovarian or cervical cancer.
5. Treatment with recombinant human granulocyte colony-stimulating factor within 6 weeks prior to enrollment.
6. Psychiatric illness or brain metastases.
7. Clinical, electrocardiographic, or other diagnostic evidence of acute congestive heart failure, cardiomyopathy, or myocardial infarction.
8. Diseases associated with splenomegaly.
9. Diagnosis of acute infection, chronic active hepatitis B within 1 year (unless known negative for hepatitis B virus antigen prior to enrollment), or hepatitis C.
10. Allergy to recombinant human granulocyte colony-stimulating factor or excipients of the study drug, or allergy to rubber.
11. Known positive serum reaction for human immunodeficiency virus (HIV) or AIDS.
12. Active tuberculosis or recent history of contact with a tuberculosis patient unless negative on tuberculin skin test, or receiving treatment for tuberculosis, or suspected case on chest X-ray examination.
13. Sickle cell anemia patients.
14. Use of other investigational drugs within 1 month prior to enrollment.
15. Patients who abuse alcohol or drugs, affecting their compliance with the study.
16. The investigator believes that the patient has a disease or symptom that makes them unsuitable for participation in this study, or that the study drug may harm the patient's health or affect the assessment of adverse events.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3/4 neutropenia | At the first of cycle 1 (each cycle is 21 days)
  Incidence of grade 3/4 neutropenia during the first chemotherapy cycle for participants receiving primary prophylaxis with Efgbemalenograstim alfa in the first treatment cycle

SECONDARY OUTCOMES:
The incidence rate of Grade 3/4 ANC reduction for each cycle | in every treatment cycle( each cycle is 21 days)
  The incidence rate of Grade 3/4 ANC reduction in every treatment cycle
The incidence rate of Grade ≥2 ANC reduction for each cycle | in every treatment cycle( each cycle is 21 days)
  The incidence rate of Grade ≥2 ANC reduction in every treatment cycle
The incidence rate of FN | in every treatment cycle( each cycle is 21 days)
  The incidence rate of febrile neutropenia (FN) for each cycle
Adverse Events | in every treatment cycle( each cycle is 21 days)
  Including adverse events/serious adverse events and their incidence rates

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Xiangya Hospital, Central South University,, Changsha, Hunan
  - Zhongda Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Qingdao Central Hospital, The Second Affiliated Hospital of Medical College of Qingdao University,, Qingdao, Shandong
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Date will be available within 6 months of study completion
Access Criteria: Date access requests will be reviewed by an external independent Review Panel.Requestors will be required to sign a Data Access Agreement.
URL: http://www.cttq.com/